CLINICAL TRIAL: NCT00107692
Title: Effect of a Weight Management Program for Overweight and Obese Children: a Randomized Controlled Trial
Brief Title: Can a Physical Activity Skill Development and Parent-Centered Dietary Intervention Help Combat Child Obesity?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Wollongong (Other)
Collaborators: Newcastle University (Other); University of Sydney (Other); Illawarra Area Health Services (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHMRC Project Grant 354101
Record Dates: First submitted 2005-04-06; First posted 2005-04-07 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2006-09

CONDITIONS: Obesity
Keywords: Child Obesity; Physical activity; community intervention study; competence; diet and nutrition; Nutrition
MeSH Terms: conditions — Obesity; Pediatric Obesity; Motor Activity | interventions — Exercise; Diet

INTERVENTIONS:
Behavioral: Physical activity and diet

SUMMARY:
The purpose of this study, and its original contribution to research, is to determine the impact of a physical activity skill development and parent centered family weight management program on the weight, cardiovascular health, physical activity, dietary intake and sedentary behaviors of overweight and obese children.

DETAILED DESCRIPTION:
AIMS

The aim of this randomized controlled trial (RCT) is to evaluate and compare in overweight children the effectiveness of the following interventions:

1. a parent-centered dietary modification program; 2. a physical activity skill development program; and 3. a parent-centered dietary modification + physical activity skill development program.

BACKGROUND

We have successfully piloted two community-based conventional weight management programs, SHARK (a physical activity-based program) and PRAISE (a dietary modification program), suitable for use with overweight, pre-adolescent children, and propose that the combination of these two programs into a multi-component intervention has the potential to effectively treat child obesity. We hypothesize that at 6-, 12-, and 24-month follow-ups, compared to overweight children allocated to the physical activity only and dietary modification only groups, overweight children in the physical activity + dietary modification group will display a greater reduction in their adiposity and display improved metabolic profiles. Secondary analyses will determine if the combined intervention improves physical activity, sedentariness, energy intake, movement skills, self-esteem, and an activity of daily living.

RESEARCH PLAN

Study design: An assessor-blinded randomized controlled trial.

Participants and their recruitment: 216 overweight children in Wollongong and Newcastle aged 6-9 years will be recruited. Each site will recruit 108 participants, 36 in each treatment arm. Recruitment will occur through the Media Units at both universities, through local GPs (general practitioners) and pediatricians.

Inclusion criteria: BMI (Body Mass Index) above international cut-off points for age and gender, one parent able to attend all required sessions, pre-pubertal, and no sibling enrolled.

Exclusion criteria: Extreme obesity (BMI SD [mean] score > 3.5), known syndromal causes of obesity, long term oral steroids, medications associated with weight gain, chronic illness, dietary restriction.

Allocation to groups: Computer-based random number-producing algorithm schedule.

Interventions: SHARK Physical activity skill development program. The "SHARK" program focuses on increasing the children's actual competence (or fundamental movement skills), perceived competence, and social support for physical activity. PRAISE parent-centered family weight management program. The PRAISE Program is a non-diet approach to healthy eating that aims to decrease overly restrictive eating and encourage eating in response to "true hunger".

Assessment of outcome variables: assessed at baseline, 6-, 12-, and 24-month follow-ups.

Adiposity: BMI SD score, height, weight, and waist circumference. Metabolic profile measures: blood pressure; cholesterol, triglycerides; glucose and insulin.

Physical activity energy expenditure and sedentary activities: total kilocalories expended and time spent in sedentary activities.

Dietary energy intake: 4-day weighed food record (2 week days and the week-end), parent selection of lower fat items in the household grocery shopping and behavior changes related to a healthy lifestyle.

Actual and perceived competence: Test of Gross Motor Development and the Self-Perception Profile for Children.

Activity of daily living: Sit-to-stand transfer.

Statistical analyses: intention-to-treat analysis using the 12-month follow-up as the initial endpoint and 24-month follow-up as final data point.

Quality-assurance. Site bias, standardized and clearly defined protocols and retention strategies have been fully addressed.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese children with the Wollongong and Newcastle regions, aged between 5.5 and 9
* BMI within specified range
* Otherwise healthy children
* Not on any medications that may influence obesity
* One parent able to attend all required sessions
* Pre-pubertal
* No sibling enrolled

Exclusion Criteria:

* Children with BMI outside the specified range
* Children on medication that may influence obesity
* Children that have conditions that may influence obesity

Ages: 66 Months to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 216
Dates: Start 2005-03; Study Completion 2007-10

PRIMARY OUTCOMES:
To evaluate and compare in overweight children the effectiveness of the following interventions: a parent-centered dietary modification program
a physical activity skill development program
and a parent-centered dietary modification + physical activity skill development program.

CONTACTS AND LOCATIONS:
Overall Officials: Tony D Okely, PhD, BEd, Principal Investigator — University of Wollongong
Locations (2):
- Australia (2):
  - University of Newcastle, Newcastle, New South Wales
  - Child Obesity Research Centre, University of Wollongong, Wollongong, New South Wales

REFERENCES:
- [Derived] Burrows T, Janet WM, Collins CE. Long-term changes in food consumption trends in overweight children in the HIKCUPS intervention. J Pediatr Gastroenterol Nutr. 2011 Nov;53(5):543-7. doi: 10.1097/MPG.0b013e3182274829. PMID 21670711
- [Derived] Collins CE, Okely AD, Morgan PJ, Jones RA, Burrows TL, Cliff DP, Colyvas K, Warren JM, Steele JR, Baur LA. Parent diet modification, child activity, or both in obese children: an RCT. Pediatrics. 2011 Apr;127(4):619-27. doi: 10.1542/peds.2010-1518. Epub 2011 Mar 28. PMID 21444600
- [Derived] Burrows T, Collins CE, Garg ML. Omega-3 index, obesity and insulin resistance in children. Int J Pediatr Obes. 2011 Jun;6(2-2):e532-9. doi: 10.3109/17477166.2010.549489. Epub 2011 Jan 12. PMID 21226540
- [Derived] Cliff DP, Okely AD, Morgan PJ, Steele JR, Jones RA, Colyvas K, Baur LA. Movement skills and physical activity in obese children: randomized controlled trial. Med Sci Sports Exerc. 2011 Jan;43(1):90-100. doi: 10.1249/MSS.0b013e3181e741e8. PMID 20473216
- [Derived] Okely AD, Collins CE, Morgan PJ, Jones RA, Warren JM, Cliff DP, Burrows TL, Colyvas K, Steele JR, Baur LA. Multi-site randomized controlled trial of a child-centered physical activity program, a parent-centered dietary-modification program, or both in overweight children: the HIKCUPS study. J Pediatr. 2010 Sep;157(3):388-94, 394.e1. doi: 10.1016/j.jpeds.2010.03.028. Epub 2010 May 6. PMID 20447648
- [Derived] Burrows T, Warren JM, Collins CE. The impact of a child obesity treatment intervention on parent child-feeding practices. Int J Pediatr Obes. 2010;5(1):43-50. doi: 10.3109/17477160902957158. PMID 19437180
- [Derived] Jones RA, Warren JM, Okely AD, Collins CE, Morgan PJ, Cliff DP, Burrows T, Cleary J, Baur LA. Process evaluation of the Hunter Illawarra Kids Challenge Using Parent Support study: a multisite randomized controlled trial for the management of child obesity. Health Promot Pract. 2010 Nov;11(6):917-27. doi: 10.1177/1524839908328994. Epub 2009 Jan 21. PMID 19158237
- [Derived] Burrows TL, Warren JM, Colyvas K, Garg ML, Collins CE. Validation of overweight children's fruit and vegetable intake using plasma carotenoids. Obesity (Silver Spring). 2009 Jan;17(1):162-8. doi: 10.1038/oby.2008.495. Epub 2008 Nov 6. PMID 18997681